CLINICAL TRIAL: NCT02156973
Title: Using Media to Reduce Anxiety for Cardiac Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14/P/059; 14/WA/0176 (Other: National Research Ethics Service)
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Anxiety
Keywords: cardiac computed tomography; Image quality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group One Usual care (No Intervention): Patients attending for CT coronary angiography all receive an information leaflet with their appointment letter, and a brief verbal description of the scan by the radiographer immediately before it is undertaken, as standard care. All patients attending will be offered the opportunity to complete a short questionnaire (until all patients are recruited - anticipated to be 4 weeks). The Speilberger State-Trait Anxiety Index has been abbreviated and validated for use in outpatient settings to gauge levels of pre-procedural anxiety. This will be undertaken on arrival and repeated immediately before the scan, to see if patients feel better prepared after the standard interaction with staff.
- Group Two Video information (Experimental): The patient video will be introduced to Group Two once Group One has been completed. In addition to the information sheet these patients (again, for four weeks or until recruitment is complete) will be sent an internet hyperlink to its presence on YouTube (video-sharing website) and the Hospital website with their appointment letter. Patients who do not have internet access will be offered the opportunity to see the video in the preparation room while waiting for their scan. Questionnaires will be administered as before, again done twice to examine any late impact of the information on patient anxiety, and the patient will undergo their test.
  Interventions: Other: Video information

INTERVENTIONS:
Other: Video information — A six minute information film to address the common themes raised by patients. This will clearly show the scanner, discuss the use of beta-blockers and radiation, and explain the likely side effects of x-ray dye (which can be alarming if patients are not expecting them). In this way we hope patients will be better prepared for the scan.
  Arms: Group Two Video information

SUMMARY:
Coming for a cardiac test can be a daunting experience. Despite providing written information sheets for patients, experience in the scanner demonstrates that many patients are ill-prepared when they attend for cardiac computed tomography (CT). Heart rate control is essential for high image quality, as this prolongs cardiac diastole (during which imaging occurs) and results in less motion blur, but this may be challenging to achieve in the context of an anxious patient. In such situations, additional radiation exposure is required to optimise the chances of diagnostic images. Thus, poor patient selection and preparation has been shown to increase the radiation burden to the patient, as well as to increase the rate of non-diagnostic scans, leading to patients needing additional, alternative testing. This can be distressing for patients and increases downstream costs for the hospital. Poor patient awareness is also known to increase the anxiety of attending for a test.

Improved patient information and understanding has been shown to improve outcomes in a wide variety of hospital settings. Evidence from cardiac catheterisation angiography suggests that the use of alternative information formats can reduce patient anxiety and improve patient satisfaction, as well as improving their understanding of the technical requirements of a test. The latter may contribute to improved preparation - for example, patients who do not understand the requirements for cardiac CT, particularly the need for a slow heart rate, will often consume caffeine, stop their heart-slowing drugs, or even run or cycle to their appointment.

We have agreed a collaboration with Plymouth University to create patient information videos for CT. These will utilise the expertise of media students (their department also runs a commercial arm, due to the quality of their output), in conjunction with the clinical requirements and patient participation groups, to create an accessible, engaging and informative film. We wish to evaluate the impact of this method of conveying information to patients on how well they are prepared to undergo testing.

If this concept is successful, it may be of use to patients undergoing a huge range of tests or treatments across specialities. We therefore need to demonstrate the efficacy (or otherwise) of such an intervention.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over 18 years attending for CT coronary angiography during the trial period will be eligible for inclusion

Exclusion Criteria:

* Unable to provide valid, informed, written consent for any reason
* Attending for non-coronary cardiac CT
* Hospital inpatients
* Patients who have previously undergone cardiac CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Self-reported level of anxiety in patients attending for CT coronary angiography. | 4 weeks
  Speilberger State-Trait Anxiety Index has been abbreviated and validated for use in outpatient settings to gauge levels of pre-procedural anxiety and will be completed by patients on arrival in the department and just before their scan.

SECONDARY OUTCOMES:
The impact of a patient information film on the pre-scan heart rate. | 4 weeks
Patient experience of scan | 2 weeks post scan
  Ten patients, selected at random from the study population, will be contacted by telephone two weeks later and a semi-structured interview will be undertaken. Patients will be questioned about how informed they felt prior to the scan, whether the scan aligned with their preconceptions, and asked to rate their overall experience.
The impact of a patient information film on the amount of use of intravenous beta blockers. | 4 weeks
The impact of a patient information film on the diagnostic image quality. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Clayton, MBBS, Study Director — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom